CLINICAL TRIAL: NCT04854525
Title: Multicenter Retrospective Evaluation Study of Pre-reconstruction Radiotherapy's Effect on One and Two Stages Prosthetic Breast Reconstruction and on Autologous Reconstruction
Brief Title: Breast Reconstruction in Previously Irradiated Breast
Status: Completed | Type: Observational
Sponsor: Humanitas Clinical and Research Center (Other)
Collaborators: Marco Klinger (Unknown); Marta Scorsetti (Unknown); Davide Franceschini (Unknown); Emanuela Morenghi (Unknown)
Responsible Party: Principal Investigator, Andrea Lisa, Principal Investigator, Humanitas Clinical and Research Center
Other Study IDs: 49/20 b
Record Dates: First submitted 2021-03-24; First posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Mammaplasty; Radiotherapy; Complications; Breast Implant; Complications; Transplant Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- One Stage Reconstruction With pre-reconstruction Radiotherapy
  Interventions: Radiation: Pre reconstruction Radiotherapy
- Two Stage Reconstruction With pre-reconstruction Radiotherapy
  Interventions: Radiation: Pre reconstruction Radiotherapy
- Autologous Reconstruction With pre-reconstruction Radiotherapy
  Interventions: Radiation: Pre reconstruction Radiotherapy
- One Stage Reconstruction Without pre-reconstruction Radiotherapy
- Two Stage Reconstruction Without pre-reconstruction Radiotherapy
- Autologous Reconstruction Without pre-reconstruction Radiotherapy

INTERVENTIONS:
Radiation: Pre reconstruction Radiotherapy — Previous PMRT
  Groups: Autologous Reconstruction With pre-reconstruction Radiotherapy; One Stage Reconstruction With pre-reconstruction Radiotherapy; Two Stage Reconstruction With pre-reconstruction Radiotherapy

SUMMARY:
For patients with breast cancer subject to a mastectomy, preserving the morphology of the breast with immediate reconstruction is a crucial aspect to preserve the quality of life.

There are several types of breast reconstruction: prosthetic in one or two stages and autologous reconstruction.

Adjuvant radiotherapy has shown an improvement of the overall survival and of the local control for patients with positive lymph nodes. As a consequence, plastic surgeons come into contact with more patients with a history of irradiation of their breasts than ever before.

However, there are few studies with a significant number that evaluate the effect of pre-reconstruction radiotherapy on the three types of reconstruction.

The aim of this study is to compare retrospectively these three types of reconstruction techniques to evaluate the impact of breast prior irradiation on the outcome of prosthetic reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patients subjected to mastectomy and immediate reconstruction directly with prostheses, in two times and by autologue flaps (TRAM, Latissimus Dorsi Flap, DIEP and any other method)

Exclusion Criteria:

* Delayed prosthetic reconstruction

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of some Breast Units in Italy
Sampling Method: Probability Sample
Enrollment: 2150 (Actual)
Dates: Start 2020-06-06 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Reconstruction failure | 2 years
  Complication rate (as hematoma, seroma, prosthetic exposure, skin and fat necrosis) that resulted in explant (prosthetic, expander or flap)

SECONDARY OUTCOMES:
Reconstruction Complications | 2 years
  Rate of need for reintervention

CONTACTS AND LOCATIONS:
Overall Officials: Marco Klinger, Study Director — Humanitas Hospital, Italy; Davide Franceschini, Study Chair — Humanitas Hospital, Italy
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Ghazal SK, Fallowfield L, Blamey RW. Comparison of psychological aspects and patient satisfaction following breast conserving surgery, simple mastectomy and breast reconstruction. Eur J Cancer. 2000 Oct;36(15):1938-43. doi: 10.1016/s0959-8049(00)00197-0. PMID 11000574
- [Background] Cordeiro PG. Breast reconstruction after surgery for breast cancer. N Engl J Med. 2008 Oct 9;359(15):1590-601. doi: 10.1056/NEJMct0802899. No abstract available. PMID 18843123
- [Background] Recht A, Comen EA, Fine RE, Fleming GF, Hardenbergh PH, Ho AY, Hudis CA, Hwang ES, Kirshner JJ, Morrow M, Salerno KE, Sledge GW Jr, Solin LJ, Spears PA, Whelan TJ, Somerfield MR, Edge SB. Postmastectomy Radiotherapy: An American Society of Clinical Oncology, American Society for Radiation Oncology, and Society of Surgical Oncology Focused Guideline Update. Pract Radiat Oncol. 2016 Nov-Dec;6(6):e219-e234. doi: 10.1016/j.prro.2016.08.009. Epub 2016 Sep 19. PMID 27659727
- [Background] Yanko-Arzi R, Cohen MJ, Braunstein R, Kaliner E, Neuman R, Brezis M. Breast reconstruction: complication rate and tissue expander type. Aesthetic Plast Surg. 2009 Jul;33(4):489-96. doi: 10.1007/s00266-008-9192-0. Epub 2008 Jun 6. PMID 18535851
- [Background] Christante D, Pommier SJ, Diggs BS, Samuelson BT, Truong A, Marquez C, Hansen J, Naik AM, Vetto JT, Pommier RF. Using complications associated with postmastectomy radiation and immediate breast reconstruction to improve surgical decision making. Arch Surg. 2010 Sep;145(9):873-8. doi: 10.1001/archsurg.2010.170. PMID 20855758
- [Background] Berry T, Brooks S, Sydow N, Djohan R, Nutter B, Lyons J, Dietz J. Complication rates of radiation on tissue expander and autologous tissue breast reconstruction. Ann Surg Oncol. 2010 Oct;17 Suppl 3:202-10. doi: 10.1245/s10434-010-1261-3. Epub 2010 Sep 19. PMID 20853034
- [Background] Chang DW, Barnea Y, Robb GL. Effects of an autologous flap combined with an implant for breast reconstruction: an evaluation of 1000 consecutive reconstructions of previously irradiated breasts. Plast Reconstr Surg. 2008 Aug;122(2):356-362. doi: 10.1097/PRS.0b013e31817d6303. PMID 18626350
- [Background] Ascherman JA, Hanasono MM, Newman MI, Hughes DB. Implant reconstruction in breast cancer patients treated with radiation therapy. Plast Reconstr Surg. 2006 Feb;117(2):359-65. doi: 10.1097/01.prs.0000201478.64877.87. PMID 16462313
- [Background] Nahabedian MY, Tsangaris T, Momen B, Manson PN. Infectious complications following breast reconstruction with expanders and implants. Plast Reconstr Surg. 2003 Aug;112(2):467-76. doi: 10.1097/01.PRS.0000070727.02992.54. PMID 12900604
- [Background] Caviggioli F, Maione L, Klinger F, Lisa A, Klinger M. Autologous Fat Grafting Reduces Pain in Irradiated Breast: A Review of Our Experience. Stem Cells Int. 2016;2016:2527349. doi: 10.1155/2016/2527349. Epub 2015 Dec 29. PMID 26858758